CLINICAL TRIAL: NCT00666458
Title: 18-wk, International, Multi-centre, Randomized, Parallel-group, Double-Blind, Active-Controlled Phase IIIb Study to Evaluate the Efficacy and Safety of Saxagliptin in Combination With Metformin in Comparison With Sitagliptin in Combination With Metformin in Adult Patients With T2D Who Have Inadequate Glycaemic Control on Metformin Alone
Brief Title: 18-week add-on to Metformin Comparison of Saxagliptin and Sitagliptin in Adult Patients With Type 2 Diabetes (T2D)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Peter Öhman, Medical Science Director, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1680C00002; EudraCT number 2007-006095-11
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Results first posted 2010-04-15 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2010-03

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): saxagliptin add-on to metformin
  Interventions: Drug: saxagliptin
- 2 (Active Comparator): sitagliptin add-on to metformin
  Interventions: Drug: sitagliptin

INTERVENTIONS:
Drug: saxagliptin — tablet, per oral, once daily
  Other Names: Onglyza
  Arms: 1
Drug: sitagliptin — capsule, per oral, once daily
  Other Names: Januvia
  Arms: 2

SUMMARY:
Saxagliptin is a new investigational medication being developed for treatment of type 2 diabetes. This study is designed to assess the efficacy and tolerability of saxagliptin in addition to metformin and compare to sitagliptin in addition with metformin.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes
* Treatment with metformin alone on stable doses of 1500 mg or higher per day for at least 8 weeks

Exclusion Criteria:

* Type 1 diabetes, history of diabetic ketoacidosis or hyperosmolar non-ketotic coma
* Insulin therapy within one year
* Previous treatment with DPP-4 inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 822 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: André Scheen, Professor, Principal Investigator — Clinical Pharmacology Unit, Liege, Belgium; Peter Öhman, MD, PhD, Study Director — AstraZeneca, Wilmington, USA; Deborah Price, MSc, Study Chair — AstraZeneca, Wilmington, USA
Locations (87):
- Argentina (9):
  - Research Site, Buenos Aires, Buenos Aires
  - Research Site, Lanús, Buenos Aires
  - Research Site, Mar del Plata, Buenos Aires
  - Research Site, Santa Fe, Santa Fe Province
  - Research Site, Caba
  - Research Site, Capital Federal
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, Rosario
- Belgium (11):
  - Research Site, Aalst, Belgium
  - Research Site, Bonheiden, Belgium
  - Research Site, Genk, Belgium
  - Research Site, Gozée, Belgium
  - Research Site, Hasselt, Belgium
  - Research Site, Liège, Belgium
  - Research Site, Saint-Médard, Belgium
  - Research Site, Sint-Gillis-Waas, Belgium
  - Research Site, Tessenderlo, Belgium
  - Research Site, Thuillies, Belgium
  - Research Site, Bruges
- Denmark (9):
  - Research Site, Aalborg
  - Research Site, Aarhus
  - Research Site, Christiansfeld
  - Research Site, Farsø
  - Research Site, Gentofte Municipality
  - Research Site, Hobro
  - Research Site, Kolding
  - Research Site, Rødovre Municipality
  - Research Site, Viborg
- France (11):
  - Research Site, Angers
  - Research Site, Château-Gontier
  - Research Site, Corbeil-Essonnes
  - Research Site, La Seyne-sur-Mer
  - Research Site, Laval
  - Research Site, Le Lavandou
  - Research Site, Montrevault
  - Research Site, Saint-Cyr
  - Research Site, Tiercé
  - Research Site, Toulon
  - Research Site, Witry-lès-Reims
- Italy (10):
  - Research Site, Bergamo, BG
  - Research Site, Foggia, FG
  - Research Site, Chiavari, GE
  - Research Site, Genova, GE
  - Research Site, Rozzano, MI
  - Research Site, Olbia, OT
  - Research Site, Padua, PD
  - Research Site, Pordenone, PN
  - Research Site, Mercato San Severino, SA
  - Research Site, Siena, SI
- Mexico (3):
  - Research Site, México, D.f.
  - Research Site, Guadalajara, Jalisco
  - Research Site, Monterrey
- Norway (10):
  - Research Site, Ålesund
  - Research Site, Elverum
  - Research Site, Halden
  - Research Site, Hamar
  - Research Site, Lierskogen
  - Research Site, Lillehammer
  - Research Site, Oslo
  - Research Site, Sandvika
  - Research Site, Strømmen
  - Research Site, Svelvik
- South Africa (10):
  - Research Site, Benoni, Gauteng
  - Research Site, Johannesburg, Gauteng
  - Research Site, Cape Town, South Africa
  - Research Site, Durban, South Africa
  - Research Site, Cape Town, Western Cape
  - Research Site, Bloemfontein
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, Kwa Zulu Natal
  - Research Site, Pretoria
- Sweden (14):
  - Research Site, Borås
  - Research Site, Degeberga
  - Research Site, Finspång
  - Research Site, Gothenburg
  - Research Site, Jönköping
  - Research Site, Ödeshög
  - Research Site, Örebro
  - Research Site, Piteå
  - Research Site, Rättvik
  - Research Site, Skanör
  - Research Site, Timrå
  - Research Site, Trollhättan
  - Research Site, Uddevalla
  - Research Site, Umeå

RESULTS

PARTICIPANT FLOW:
Groups:
- Saxa + Met: Saxagliptin 5 mg tablets added on to open-label metformin
- Sita + Met: Sitagliptin 100 mg capsules added on to open-label metformin
Period: Overall Study
Arm/Group | Saxa + Met | Sita + Met
Started | 403 (Randomized and treated) | 398 (Randomized and treated)
Completed | 365 (Completed 18 weeks of treatment) | 374 (Completed 18 weeks of treatment)
Not Completed | 38 | 24
Not completed — Adverse Event | 8 | 7
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Lost to Follow-up | 0 | 3
Not completed — Administrative reason by sponsor | 1 | 1
Not completed — Incorrect enrollment | 7 | 1
Not completed — Study specific discontinuation criteria | 14 | 7
Not completed — Severe non-compliance to the protocol | 1 | 1
Not completed — Safety reasons | 1 | 0
Not completed — Medical history of anemia | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxa + Met | Sita + Met | Total
Number analyzed (Participants) | 403 | 398 | 801
Age Continuous [Mean (Standard Deviation); unit: years] | 58.77 (10.14) | 58.07 (10.51) | 58.42 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 213 | 196 | 409
  Male | 190 | 202 | 392

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c (HbA1c) Change From Baseline to Week 18
Description: Adjusted mean change from baseline in HbA1c achieved with saxagliptin added on to metformin versus sitagliptin added on to metformin at Week 18 (Per Protocol Analysis Set). HbA1c is a continuous measure, the change from baseline for each participant is calculated as the Week 18 value minus the baseline value.
Time Frame: Baseline, Week 18
Population: Randomized participants who completed the 18 weeks of treatment had both baseline and week 18 HbA1c measurement and had no significant protocol deviations.
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Saxa + Met | Sita + Met
Number analyzed (Participants) | 334 | 343
Percent
  Baseline | 7.68 (0.052) | 7.69 (0.047)
  Week 18 | 7.16 (0.052) | 7.07 (0.051)
  Adjusted Change from Baseline | -0.52 (0.039) | -0.62 (0.038)
Statistical Analysis 1: Comparison: Saxa + Met vs Sita + Met; Test type: Superiority or Other; Mean Difference (Net) = 0.09, 95% CI 2-sided [-0.01 to 0.20], Standard Error of Mean 0.055

2. Secondary Outcome: Proportion of Patients Achieving Therapeutic Glycaemic Response Defined as HbA1c <= 6.5% at Week 18
Description: Proportion of Patients Achieving Therapeutic Glycaemic Response Defined as HbA1c <= 6.5% at Week 18 (Full Analysis Set)
Time Frame: Week 18 (Last Observation Carried Forward)
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in the Week 18 LOCF analysis, participants must have had a baseline and at least 1 post-baseline measurement.
Measure: Number; unit: Percentage of Participants
Arm/Group | Saxa + Met | Sita + Met
Number analyzed (Participants) | 399 | 392
Percentage of Participants | 26.3 | 29.1
Statistical Analysis 1: Comparison: Saxa + Met vs Sita + Met; Test type: Superiority or Other; Difference in Percent = -2.8, 95% CI 2-sided [-9.0 to 3.5]

3. Secondary Outcome: Fasting Plasma Glucose Change From Baseline to Week 18 (mg/dL)
Description: Adjusted mean change from baseline in Fasting Plasma Glucose achieved with saxagliptin added on to metformin versus sitagliptin added on to metformin at Week 18 (Full Analysis Set). Fasting Plasma Glucose is a continuous measure, the change from baseline for each participant is calculated as the Week 18 (LOCF) value minus the baseline value.
Time Frame: Baseline, Week 18 (Last Observation Carried Forward)
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in analysis of change from baseline to Week 18 LOCF, participants must have had a baseline and at least 1 post-baseline measurement.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxa + Met | Sita + Met
Number analyzed (Participants) | 397 | 392
mg/dL
  Baseline | 159.67 (2.280) | 160.22 (2.192)
  Week 18 | 149.04 (1.991) | 143.94 (1.864)
  Adjusted Change from Baseline | -10.75 (1.455) | -16.16 (1.464)
Statistical Analysis 1: Comparison: Saxa + Met vs Sita + Met; Test type: Superiority or Other; Mean Difference (Net) = 5.42, 95% CI 2-sided [1.37 to 9.47], Standard Error of Mean 2.064

4. Secondary Outcome: Fasting Plasma Glucose Change From Baseline to Week 18 (mmol/L)
Description: as for outcome 3
Time Frame: Baseline, Week 18 (Last Observation Carried Forward)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Saxa + Met | Sita + Met
Number analyzed (Participants) | 397 | 392
mmol/L
  Baseline | 8.86 (0.127) | 8.89 (0.122)
  Week 18 | 8.27 (0.111) | 7.99 (0.103)
  Adjusted Change from Baseline | -0.60 (0.081) | -0.90 (0.081)
Statistical Analysis 1: Comparison: Saxa + Met vs Sita + Met; Test type: Superiority or Other; Mean Difference (Net) = 0.30, 95% CI 2-sided [0.08 to 0.53], Standard Error of Mean 0.115

ADVERSE EVENTS:
Arm/Group | Saxa + Met | Sita + Met
Serious Adverse Events (participants affected / at risk) | 7/403 | 5/398
Other Adverse Events (participants affected / at risk) | 54/403 | 50/398
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saxa + Met (N=403) | Sita + Met (N=398)
Chills (General disorders) | 1 | 0
Ulcer Haemorrhage (General disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemic Unconsciousness (Metabolism and nutrition disorders) | 0 | 1
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saxa + Met (N=403) | Sita + Met (N=398)
Urinary Tract Infection (Infections and infestations) | 28 | 26
Influenza (Infections and infestations) | 27 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No